CLINICAL TRIAL: NCT02591979
Title: PASHOS Project: Advanced Platform for Sleep Apnea Syndrome Assessment. A Multi-Centre Study to Validate a Sleep Apnea Screening Model in Primary Health Care
Brief Title: PASHOS Project: Advanced Platform for Sleep Apnea Syndrome Assessment
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-PAS-2013-151
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea Syndrome
Keywords: Sleep Apnea Syndrome; Primary Health Care
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop and validate a work-model in Primary Health Care for identifying patients with Sleep Apnea Syndrome, based on clinical variables and an ambulatory monitoring study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 75 years.

Exclusion Criteria:

* Cognitive impairment or psycho-physical deterioration that impede to perform ambulatory monitoring study.
* Worsened or unstable cardiovascular or cerebrovascular disease.
* Chronic insomnia (<5h sleep / day).
* Relevant respiratory comorbidity that could interfere with arterial saturation measurements, as moderate to severe chronic obstructive pulmonary disease.
* Neuromuscular disease.
* Refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visited at Primary Care consultations will be included according to a randomization schedule to reach the necessary sample.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Apnea/Hypopnea Index | At baseline
  At primary healthcare
Apnea/Hypopnea Index | At 3 months
  At Sleep Lab Unit

SECONDARY OUTCOMES:
Cardiovascular risk factors | At baseline
History of cardiovascular or cerebrovascular disease | At baseline
Lung function tests | At baseline
Self-perceived sleepiness. Epworth Test | At baseline
  At primary healthcare
Self-perceived sleepiness. Epworth Test | At 3 months
  At Sleep lab unit

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Penacoba P, Llauger MA, Fortuna AM, Flor X, Sampol G, Pedro-Pijoan AM, Grau N, Santiveri C, Juvanteny J, Aoiz JI, Bayo J, Lloberes P, Mayos M; PASHOS Working Group. A new tool to screen patients with severe obstructive sleep apnea in the primary care setting: a prospective multicenter study. BMC Pulm Med. 2022 Jan 15;22(1):38. doi: 10.1186/s12890-022-01827-0. PMID 35033055
- [Derived] Penacoba P, Llauger MA, Fortuna AM, Flor X, Sampol G, Pedro Pijoan AM, Grau N, Santiveri C, Juvanteny J, Aoiz JI, Bayo J, Lloberes P, Mayos M; PASHOS Working Group. Primary care and sleep unit agreement in management decisions for sleep apnea: a prospective study in Spain. J Clin Sleep Med. 2020 Sep 15;16(9):1579-1589. doi: 10.5664/jcsm.8492. PMID 32279702